CLINICAL TRIAL: NCT03985540
Title: Treating Cognitive Deficits in Traumatic Spinal Cord Injury (SCI): A Randomized Clinical Trial
Brief Title: Treating Cognitive Deficits in Traumatic Spinal Cord Injury (SCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nancy Chiaravalloti, Director NNL & TBI, Kessler Foundation
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: R-947-16
Record Dates: First submitted 2017-08-15; First posted 2019-06-13 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- memory experimental group (Experimental): Experimental group will receive memory retraining exercises administered on a lab top computer twice a week for 5 weeks.
  Interventions: Behavioral: Behavorial; memory exercise
- Placebo comparator memory (Placebo Comparator): Placebo controlled group will receive placebo memory retraining exercises administered on a lab top computer twice a week for 5 weeks.
  Interventions: Behavioral: Placebo; memory exercise
- Processing speed (Experimental): Processing speed group will receive processing speed training exercises administered on a lab top computer twice a week for 5 weeks.
  Interventions: Behavioral: Behavioral: speed exercises
- Processing speed placebo (Placebo Comparator): Placebo controlled group will receive placebo processing speed training exercises administered on a lab top computer twice a week for 5 weeks.
  Interventions: Behavioral: Placebo speed training

INTERVENTIONS:
Behavioral: Behavorial; memory exercise — Memory training twice a week for 5 weeks.
  Arms: memory experimental group
Behavioral: Placebo; memory exercise — Placebo Memory training twice a week for 5 weeks
  Arms: Placebo comparator memory
Behavioral: Behavioral: speed exercises — Speed training twice a week for 5 weeks.
  Arms: Processing speed
Behavioral: Placebo speed training — Placebo Speed training twice a week for 5 weeks.
  Arms: Processing speed placebo

SUMMARY:
The purpose of this research study is to investigate the effectiveness of a memory retraining program and a processing speed program in a spinal cord injured (SCI) population. The study is designed to research how well different types of techniques can help people with SCI improve in areas where they might have difficulties such as memory or processing speed, (time it takes to process information provided).

DETAILED DESCRIPTION:
The objectives of the currently proposed randomized clinical trial are to (1) apply a treatment protocol for Processing Speed and Learning and memory impairments, well-validated in other neurological populations, to individuals with SCI with objectively observable deficits in these areas and document efficacy on standard neuropsychological testing; (2) assess the effectiveness of the interventions in persons with SCI utilizing global measures of everyday life; (3) evaluate the long-term benefit of treatment. Prior to enrollment in the study protocol, all potential subjects will undergo a 2-part screening: (1) an initial screening examination via telephone during which basic information will be gathered and (2) a detailed, in-person screening that will be completed on if the subject passes the initial screen. Individuals must meet full screening criteria to be eligible for participation.

ELIGIBILITY:
Inclusion Criteria:

* I am between the ages of 18 and 75 years old.
* I have a spinal cord injury with the level of injury between C1-T12.
* I am non-ambulatory (I use a wheelchair as my primary means of getting around).
* I have an AIS grade of A, B or C as determined by study staff examination.
* My injury occurred at least 1 year ago.
* My primary language is English.

Exclusion Criteria:

* I have a current illness or infection. My enrollment in this study can be delayed until my current illness or infection is successfully treated.
* I have any neurological condition other than SCI (Alzheimer's disease, dementia, stroke, multiple sclerosis, Parkinson's disease, etc.).
* I have a diagnosis of a psychiatric disorder such as post-traumatic stress disorder, schizophrenia or bipolar disorder.
* I have a history of Hypertension or Diabetes Mellitus (due to its impact on brain function).
* My vision is impaired- more than 20/60 in worst eye (with prescription eyewear).
* I have been taking steroids, benzodiazepines, or certain neuroleptics within past month, the study doctor will review my medications with me.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2016-11-16 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
California Verbal Learning Test | Assessments will look at change over 6 weeks of treatment and 3 months after completion
  California Verbal Learning TestPerformance on a memory test using the

SECONDARY OUTCOMES:
SCI Quality of Life Scale | Assessments will look at change over 6 weeks of treatment and 3 months after completion
  Reports on emotional functioning, memory functioning and quality of life using the SCI Quality of Life Scale, which measures all of these constructs. DVs will be the depression subscale (range: 0-40; lower score is better) and cognitive subscale (range:0-40; higher score is better).

OTHER OUTCOMES:
Symbol-Digit Modalities Test (oral form) | Assessments will look at change over 6 weeks of treatment and 3 months after completion
  Performance on processing speed test, Symbol-Digit Modalities Test (oral form)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Green, PhD, Study Chair — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States